CLINICAL TRIAL: NCT04208087
Title: A Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of SI-722 Intravesical Instillation in Interstitial Cystitis/Bladder Pain Syndrome Subjects
Brief Title: PK and Safety of SI-722 in IC/BPS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Seikagaku Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 722/1121
Record Dates: First submitted 2019-11-25; First posted 2019-12-23 (Actual); Results first posted 2023-12-29 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Interstitial Cystitis; Bladder Pain Syndrome
Keywords: Bladder; Intravesical Injection; Interstitial Cystitis
MeSH Terms: conditions — Cystitis, Interstitial

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SI-722 (Experimental)
  Interventions: Drug: SI-722
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SI-722 — SI-722 will be intravesically instilled.
  Arms: SI-722
Drug: Placebo — Placebo will be intravesically instilled.
  Arms: Placebo

SUMMARY:
This study is designed randomized, double-blind, placebo-controlled trial in Interstitial Cystitis/Bladder Pain Syndrome patients.

ELIGIBILITY:
Inclusion Criteria:

* Males or females, ≥18 and ≤80 years of age
* A score of 19 or greater on the Bladder Pain/Interstitial Cystitis Symptom Score (BPIC-SS)

Exclusion Criteria:

* Urinary tract infection ≤30 days
* Treatment with intravesical therapy ≤60 days
* Treatment with any opioid therapy ≤7 days
* History of bladder hydrodistension ≤3 months
* Has cancer or a past history of any cancer ≤5 years
* Body mass index (BMI) ≥40 kg/m2

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2020-03-30 (Actual); Primary Completion 2021-01-12 (Actual); Study Completion 2021-01-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - American Institute of Research, Los Angeles, California
  - TriValley Urology Medical Group, Murrieta, California
  - Premier Medical Associates, The Villages, Florida
  - AccuMed Research Associates, Garden City, New York
  - Centex Studies, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: The participants received a single intravesical instillation of Placebo
- Low Dose of SI-722: The participants received a single intravesical instillation of Low Dose of SI-722
- Medium Dose of SI-722: The participants received a single intravesical instillation of Medium Dose of SI-722
- Medium-high Dose of SI-722: The participants received a single intravesical instillation of Medium-high Dose of SI-722
- High Dose of SI-722: The participants received a single intravesical instillation of High Dose of SI-722
Period: Overall Study
Arm/Group | Placebo | Low Dose of SI-722 | Medium Dose of SI-722 | Medium-high Dose of SI-722 | High Dose of SI-722
Started | 8 | 6 | 6 | 6 | 7
Completed | 7 | 6 | 5 | 6 | 6
Not Completed | 1 | 0 | 1 | 0 | 1
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Low Dose of SI-722 | Medium Dose of SI-722 | Medium-high Dose of SI-722 | High Dose of SI-722 | Total
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 7 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.6 (16.15) | 41.8 (6.40) | 51.0 (14.91) | 54.0 (17.79) | 45.4 (11.47) | 49.8 (14.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 5 | 4 | 7 | 25
  Male | 2 | 3 | 1 | 2 | 0 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 5 | 3 | 1 | 1 | 12
  Not Hispanic or Latino | 6 | 1 | 3 | 5 | 6 | 21
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 0 | 0 | 2 | 5
  White | 6 | 5 | 5 | 6 | 5 | 27
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Body Mass Index [Mean (Standard Deviation); unit: kilograms/meter square] | 27.13 (5.79) | 32.52 (4.37) | 26.20 (3.23) | 23.63 (3.39) | 28.59 (6.01) | 27.61 (5.35)

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax) for SI-722
Description: SI-722 concentrations in plasma were measured using collected blood samples, and plasma PK parameters for SI-722 were estimated.
Time Frame: 4 weeks
Population: The PK Population is defined as all subjects who received SI-722 and who provided at least 1 evaluable PK sample. One participant in the High Dose group was excluded from PK population because the subject discontinued before IP administration due to difficulty with drawing blood.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Low Dose of SI-722 | Medium Dose of SI-722 | Medium-high Dose of SI-722 | High Dose of SI-722
Number analyzed (Participants) | 6 | 6 | 6 | 6
ng/mL | NA (NA) — Plasma PK parameters of SI-722 were not calculated because the plasma SI-722 concentrations were BLQ in all subjects. | NA (NA) — Plasma PK parameters of SI-722 were not calculated because the plasma SI-722 concentrations were BLQ in all subjects. | NA (NA) — Plasma PK parameters of SI-722 were not calculated because the plasma SI-722 concentrations were BLQ in all subjects. | NA (NA) — Plasma PK parameters of SI-722 were not calculated because the plasma SI-722 concentrations were BLQ in all subjects.

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Placebo | Low Dose of SI-722 | Medium Dose of SI-722 | Medium-high Dose of SI-722 | High Dose of SI-722
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/6 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 4/8 | 1/6 | 1/6 | 3/6 | 3/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=8) | Low Dose of SI-722 (N=6) | Medium Dose of SI-722 (N=6) | Medium-high Dose of SI-722 (N=6) | High Dose of SI-722 (N=6)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Genital herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-17): https://cdn.clinicaltrials.gov/large-docs/87/NCT04208087/Prot_SAP_000.pdf